CLINICAL TRIAL: NCT07384793
Title: Comparison of Efficacy of Azithromycin Alone vs Combination of Azithromycin and Probiotics in Management of Mild to Moderate Acne Vulgaris
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hayatabad Medical Complex (Other Government)
Responsible Party: Principal Investigator, Naheed asghar, Associate Professor Dermatology unit HMC, Hayatabad Medical Complex
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMC Peshawar
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-10

CONDITIONS: Acne Vulgaris II or III Degree
MeSH Terms: interventions — Azithromycin; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Azithromycin group (Active Comparator): The participants in this arm of study will receive only Oral Azithromycin to treat their Acne
  Interventions: Drug: Azithromycin 250 MG Oral Capsule
- Oral Azithromycin and Oral probiotic combination (Active Comparator): The participants in this arm of study will receive both Oral Azithromycin and Oral Probiotics to treat their Acne
  Interventions: Drug: Azithromycin 250 MG Oral Capsule Along with Oral Probiotics

INTERVENTIONS:
Drug: Azithromycin 250 MG Oral Capsule — The participants in this arm of study will receive only Oral Azithromycin 250mg on alternate day for 12 weeks to treat their Acne
  Arms: Oral Azithromycin group
Drug: Azithromycin 250 MG Oral Capsule Along with Oral Probiotics — The participants in this arm of study will receive only Oral Azithromycin 250mg on alternate day along with oral probiotics daily for 12 weeks to treat their Acne
  Arms: Oral Azithromycin and Oral probiotic combination

SUMMARY:
The Goal of this Clinical trial is to compare the efficacy of oral azithromycin alone with combination therapy of oral azithromycin and probiotics to see is there any significant difference in outcome of two treatment modalities in mild to moderate acne vulgaris

ELIGIBILITY:
Inclusion Criteria: Participants with mild to moderate acne on basis of global acne assessment scale score of 2 or 3 and with 20 to 50 total lesion count will be included.

-

Exclusion Criteria:

History of active localized or generalized infection History of autoimmune disease History of other facial skin diseases/ excessive facial hair or scars History of using isotretinoin or oral contraceptive pills in past 6 months History of already using antibiotics for acne treatment History of facial cosmetic procedures within last 3 months History of allergy to drugs used in study History of using drugs that may interact with azithromycin Currently pregnant or lactating women

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Reduction of Acne Lesion Count as per Acne Global assessment scale | 12 Weeks
  The patients will be assessed before and after the treatment and their lesions will be counted .The Primary outcome that will be measured is the reduction of the lesion counts according to the Acne global Assessment scale
  The participants included will be with mild to moderate acne on basis of global acne assessment scale score of 2 or 3.
  The minimum Lesion count considered will be 20 and the Maximum will be 50.
  Lower is better Higher is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Naeem, Study Chair — Hayatabad Medical Complex Peshawar, KPK Pakistan
Locations (1):
- Hayatabad Medical Complex, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: No